CLINICAL TRIAL: NCT06219083
Title: Study of Nutritional Status and Clinical Outcomes in Patients With Common Malignancies
Brief Title: Nutritional Status and Clinical Outcomes in Patients With Common Malignancies(NCOM)
Acronym: NCOM
Status: Recruiting | Type: Observational
Sponsor: Xiaoqin Luo (Other)
Responsible Party: Sponsor-Investigator, Xiaoqin Luo, Professor, Xi'an Jiaotong University
Organization: Xi'an Jiaotong University (Other)
Other Study IDs: 2022-1373
Record Dates: First submitted 2023-12-23; First posted 2024-01-23 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Chemoradiotherapy; Nutrition, Healthy; Oncology; Clinical Outcomes
Keywords: Chemoradiotherapy; Nutritional Status in Cancer Patients; Clinical Outcomes of Cancer Treatment; Cancer Patient Nutrition; Shaanxi Province Cancer Study
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumor tissue, paracancerous tissue, Serum, Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter, prospective cohort study investigates the long-term impact of nutritional status on clinical outcomes in cancer patients undergoing treatment in Shaanxi Province, China. It evaluates how malnutrition, dietary patterns, and nutritional interventions affect treatment tolerance, quality of life, and survival. The study tracks dynamic changes in nutritional health and related indicators throughout various stages of chemoradiotherapy, aiming to inform evidence-based strategies for precision nutrition in oncology care.

DETAILED DESCRIPTION:
Study Purpose and Objectives:

The Nutritional Status and Clinical Outcomes in Patients with Common Malignancies (NCOM) study aims to assess how nutritional status influences treatment-related complications, functional performance, psychosocial well-being, and long-term survival in cancer patients. By capturing longitudinal data, the study seeks to identify modifiable risk factors and develop predictive models to support personalized nutritional interventions in oncology.

Study Design and Scope:

The study is being conducted at 11 tertiary hospitals across Xi'an, Shaanxi Province, and will recruit a total of 1,538 patients diagnosed with common malignancies. Participants are enrolled within 48 hours of hospital admission and followed at structured intervals over a five-year period: at 1, 2, 3, 6, and 12 months, and then annually. Baseline and follow-up evaluations include demographic data, cancer-specific clinical characteristics, nutritional risk (mPG-SGA, NRS-2002), dietary intake (SDSAT), quality of life (EORTC QLQ-C30), psychosocial health (HADS), physical activity, sleep quality (PSQI), and laboratory biomarkers.

Data Collection and Management:

Standardized procedures are used for anthropometric measurements, clinical assessments, and patient-reported outcomes. Nutritional support in and out of hospital, inflammatory biomarkers, liver and kidney function, and hematological indicators are systematically recorded. All data are managed via REDCap with built-in validation, routine audits, and centralized oversight.

Quality Assurance and Training:

Research personnel at each site undergo rigorous training to ensure consistency in data collection and patient evaluation. Supervisors oversee data quality, coordinate follow-up, and address missing data or protocol deviations.

Ethical Oversight:

The study adheres to the Declaration of Helsinki and was approved by the Ethics Committee of Xi'an Jiaotong University Health Science Center (Approval No. 2022-1373). Written informed consent is obtained from all participants. All personal data are deidentified and securely stored.

Expected Outcomes and Significance:

By establishing the temporal relationships between nutritional status and clinical outcomes, the NCOM study will provide high-quality evidence to support individualized nutrition-focused care. Results are expected to improve early identification of patients at risk, optimize nutritional interventions, reduce treatment-related toxicity, and enhance long-term cancer prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above
* Pathologically diagnosed with malignant tumors
* Scheduled to undergo radiotherapy and/or chemotherapy
* Clear consciousness, no communication barriers
* Willing to undergo follow-up, not in a near-death condition

Exclusion Criteria:

* Patients without a pathological diagnosis of malignant tumors
* Patients with AIDS
* Patients with mental or cognitive disorders
* Patients who have undergone organ transplantation
* Patients with a life expectancy less than 12 months
* Pregnant women
* Patients currently participating in other clinical intervention studies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cancer patients from 20 hospitals in Shaanxi Province undergoing chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 1538 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Nutritional Status Assessed by Modified Patient-Generated Subjective Global Assessment (mPG-SGA) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Longitudinal assessment of nutritional status using the mPG-SGA, a validated tool composed of five sections (weight loss history, dietary intake, symptoms, function/activity, and age). Total scores range from 0 to ≥7 points, with higher scores indicating worse nutritional status. Patients will be classified as:
  0-2 = Normal
  3-6 = Mild malnutrition
  ≥7 = Moderate to severe malnutrition.
Change in Nutritional Risk Assessed by Nutritional Risk Screening 2002 (NRS-2002) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Longitudinal evaluation of nutritional risk using the NRS-2002, which considers disease severity, nutritional impairment, and age. Total score ranges from 0 to ≥7 points. A score of ≥3 indicates nutritional risk and warrants intervention; <3 indicates no immediate risk.
Change in Global Health Status Score on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Assessment of patients' perceived overall health status using the global health subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). Scores range from 0 to 100, with higher scores indicating better global quality of life.
Change in Functional Scores on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Evaluation of physical, role, emotional, cognitive, and social functioning domains using the functional scales of the EORTC QLQ-C30. Each domain score ranges from 0 to 100, with higher scores representing better functioning. Each domain will be reported separately.
Change in Symptom Scores on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Assessment of symptom burden including fatigue, pain, nausea/vomiting, appetite loss, sleep disturbance, constipation, diarrhea, and financial difficulty using symptom subscales of the EORTC QLQ-C30. Each symptom is scored separately from 0 to 100, with higher scores indicating worse symptom severity.
Overall Survival (OS) in Cancer Patients | From date of enrollment until death or last follow-up (up to 5 years)
  Overall survival is defined as the time from the date of enrollment to the date of death from any cause. Patients still alive at the last follow-up will be censored. Kaplan-Meier survival analysis and Cox proportional hazards regression will be used to estimate survival and explore associations with baseline and longitudinal nutritional status.
Progression-Free Survival (PFS) in Cancer Patients | From date of enrollment until death or last follow-up (up to 5 years)
  Progression-free survival is defined as the time from enrollment to the first documented disease progression or death from any cause, whichever occurs first. Patients without progression at the time of last follow-up will be censored. PFS will be analyzed using Kaplan-Meier estimates and Cox regression models, stratified by nutritional status.

SECONDARY OUTCOMES:
Serum Total Protein | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Serum total protein concentration (g/L), used to evaluate protein-energy nutritional status. Measured using standard biochemical assays.
Serum Albumin | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Serum albumin concentration (g/L), used to assess visceral protein status and systemic inflammation.
Serum Prealbumin | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Serum prealbumin level (mg/L), an indicator of short-term changes in protein-energy nutritional status.
Serum Transferrin | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Serum transferrin concentration (g/L), a marker of protein status and iron metabolism.
C-Reactive Protein (CRP) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Serum CRP (mg/L), a marker of systemic inflammation and acute-phase response.
Blood Glucose | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Fasting blood glucose (mmol/L), measured to assess metabolic function and risk of hyperglycemia.
Aspartate Aminotransferase (AST) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  AST concentration (U/L), used as a liver function test and hepatotoxicity marker.
Alanine Aminotransferase (ALT) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  ALT level (U/L), a liver enzyme measured to monitor hepatic injury.
Interleukin-1 (IL-1) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  IL-1 concentration (pg/mL), a pro-inflammatory cytokine indicative of immune and inflammatory activity.
Tumor Necrosis Factor-alpha (TNF-α) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Tumor Necrosis Factor-alpha (TNF-α) level (pg/mL) measured to assess systemic inflammation and cancer-related cachexia.
Serum Creatinine | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Serum creatinine (μmol/L), measured to evaluate kidney function and treatment-related nephrotoxicity.
Blood Urea Nitrogen | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Blood urea nitrogen (umol/L), used to monitor renal function and protein catabolism.
Total Bilirubin | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  umol/LBlood urea nitrogen (umol/L), used to monitor renal function and protein catabolism.
Direct Bilirubin | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Direct (conjugated) bilirubin (μmol/L), used to evaluate biliary obstruction and liver function.
Total Cholesterol | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Total cholesterol level (mmol/L), measured to assess lipid metabolism and nutritional status.
Triglycerides | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Serum triglyceride level (mmol/L), used to evaluate energy reserves and lipid metabolism.
High-Density Lipoprotein Cholesterol (HDL-C) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  HDL-C (mmol/L), assessed as a marker of cardiovascular health and lipid status.
Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  LDL-C (mmol/L), measured as a risk factor for cardiovascular disease and lipid status.
Interleukin-6 (IL-6) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  IL-6 level (pg/mL), a pro-inflammatory cytokine measured to monitor systemic inflammation and cachexia.
Hemoglobin | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Hemoglobin concentration (*10⁹/L), used to assess anemia and oxygen-carrying capacity.
White Blood Cell Count (Leukocytes) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Total white blood cell count (*10⁹/L), measured to monitor immune status and detect infection or myelosuppression.
Neutrophil Count | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Absolute neutrophil count (*10⁹/L), used to assess infection risk and bone marrow suppression.
Lymphocyte Count | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Lymphocyte count (*10⁹/L), measured to evaluate immune competence.
Red Blood Cell Count | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Red blood cell count (*10¹²/L), used to assess erythropoiesis and anemia.
Platelet Count | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Platelet count (*10⁹/L), measured to evaluate coagulation status and myelosuppression.
Height | through study completion, an average of 1 year
  Standing height (cm) measured using a stadiometer with 0.5 cm precision. Values adjusted for presence of ascites, edema, or large tumors.ascites, systemic edema, and huge tumors.
Body Weight | through study completion, an average of 1 year
  Body weight (kg) measured using a calibrated scale with 0.2 kg precision. Values adjusted if ascites or edema are present.
Body Mass Index (BMI) | through study completion, an average of 1 year
  BMI calculated as weight (kg) divided by height squared (m²), recorded to one decimal place.
Change in Anxiety Symptoms Assessed by Hospital Anxiety and Depression Scale (HADS-A) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Change in Anxiety Symptoms Assessed by Hospital Anxiety and Depression Scale (HADS-A)
Change in Depression Symptoms Assessed by Hospital Anxiety and Depression Scale (HADS-D) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Assessment of depressive symptoms using the HADS-D subscale of the Hospital Anxiety and Depression Scale. Scores range from 0 to 21, with higher scores indicating more severe depression. Results will be analyzed in relation to nutritional status (normal, mild, moderate malnutrition).
Functional Performance Measured by Karnofsky Performance Status (KPS) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Functional performance will be evaluated using the Karnofsky Performance Status (KPS) scale, which ranges from 0 to 100. Higher scores indicate better functional ability and independence in daily activities. Longitudinal KPS changes will be assessed in relation to changes in nutritional status over time.
Changes in Sleep Quality Assessed by Pittsburgh Sleep Quality Index (PSQI) | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Sleep quality and disturbances will be evaluated using the Pittsburgh Sleep Quality Index (PSQI), a standardized questionnaire assessing seven components of sleep. Total scores range from 0 to 21, with higher scores indicating poorer sleep quality. PSQI scores will be analyzed in relation to nutritional risk categories and treatment phases.
Changes in Physical Activity Level During Cancer Treatment | Baseline, 1, 2, 3, 6, and 12 months after admission; annually up to 5 years
  Assessment of leisure-time physical activity levels (mild, moderate, vigorous) and their relationship with nutritional status and cancer treatment response.
Changes in Nutrition-Related Knowledge, Attitudes, and Practices (KAP) | Baseline, 6 months, and 12 months after admission; annually up to 5 years
  Patients' dietary knowledge, attitudes, and practices will be assessed using a validated Nutrition KAP (Knowledge, Attitude, and Practice) questionnaire. The total score ranges from 0 to 104, with higher scores indicating better nutritional knowledge, more positive attitudes, and healthier dietary behaviors. Longitudinal changes in KAP scores will be evaluated in relation to treatment outcomes.
Healthcare Utilization and Cost of Nutrition-Related Care | From admission through 30-day post-discharge and annually for 5 years
  Evaluation of healthcare utilization related to nutritional care, including total number of hospitalization days, number of ICU admissions, and direct costs associated with enteral and parenteral nutrition support. Metrics will be analyzed in relation to malnutrition risk at baseline and during treatment.
Incidence of Serious Adverse Events Related to Nutrition or Treatment | Continuously from enrollment through end of study follow-up (up to 5 years)
  Tracking of serious adverse events potentially related to nutritional support or treatment, including infections, allergic reactions, gastrointestinal distress, and metabolic complications.

OTHER OUTCOMES:
Predictive Value of Baseline Nutritional Indicators for 30-Day Clinical Events | Baseline to 30 days post-admission
  Evaluation of whether baseline nutritional indicators-including mPG-SGA scores and laboratory biomarkers such as albumin, prealbumin, and CRP-predict 30-day clinical outcomes, including mortality, ICU admission, and significant unintentional weight loss (>5%). Logistic regression will be used for model construction and discrimination.
Nutritional Trajectory Typing and Clustering | From baseline to 12-month follow-up
  Identification of distinct nutritional change trajectories over time using latent class growth analysis (LCGA) and hierarchical clustering based on serial measurements of mPG-SGA and anthropometric data. Trajectories will be used to classify patients into nutritional risk subgroups.
Agreement Between Nutritional Screening Tools (mPG-SGA vs. NRS-2002) | Baseline and each scheduled follow-up visit (up to 5 years)
  Assessment of the diagnostic agreement, sensitivity, and specificity of two nutritional screening tools-modified Patient-Generated Subjective Global Assessment (mPG-SGA) and Nutritional Risk Screening 2002 (NRS-2002)-in detecting malnutrition risk. Agreement will be evaluated using Cohen's kappa and ROC curve analysis.
Sociodemographic Determinants of Malnutrition | From baseline throughout study follow-up (up to 5 years)
  Analysis of sociodemographic factors-including income level, education, employment status, and rural vs. urban residence-in predicting baseline malnutrition and nutritional deterioration over time. Multivariable models will be used to explore independent associations.
Patient Adherence to Out-of-Hospital Nutritional Support | Baseline to 12 months post-treatment initiation
  Evaluation of patient-reported adherence to prescribed oral nutritional supplements or enteral/parenteral support regimens after hospital discharge. Adherence data will be collected via structured interviews and compared with clinical outcomes and readmission rates.

CONTACTS AND LOCATIONS:
Locations (1):
- Xi 'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
The study intends to share IPD with other researchers for advancing scientific understanding and improving patient care. The shared data will include anonymized participant information, such as demographic details, clinical outcomes, and treatment responses. The data will be stripped of any identifiers to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available after the publication of the main study results, anticipated to be by the end of 2025. The data will be accessible for a period of five years following this date.
Access Criteria: Researchers interested in accessing the data will be required to submit a proposal outlining their intended use of the data, which will be reviewed by the study's principal investigator. Access will be granted based on the scientific merit and ethical considerations of the proposal.

REFERENCES:
- [Background] Baracos VE. Cancer-associated malnutrition. Eur J Clin Nutr. 2018 Sep;72(9):1255-1259. doi: 10.1038/s41430-018-0245-4. Epub 2018 Sep 5. No abstract available. PMID 30185853
- [Background] Muscaritoli M, Corsaro E, Molfino A. Awareness of Cancer-Related Malnutrition and Its Management: Analysis of the Results From a Survey Conducted Among Medical Oncologists. Front Oncol. 2021 May 13;11:682999. doi: 10.3389/fonc.2021.682999. eCollection 2021. PMID 34055649
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424
- [Result] Morgan E, Arnold M, Gini A, Lorenzoni V, Cabasag CJ, Laversanne M, Vignat J, Ferlay J, Murphy N, Bray F. Global burden of colorectal cancer in 2020 and 2040: incidence and mortality estimates from GLOBOCAN. Gut. 2023 Feb;72(2):338-344. doi: 10.1136/gutjnl-2022-327736. Epub 2022 Sep 8. PMID 36604116
- [Result] Zhou J, Zheng R, Zhang S, Zeng H, Wang S, Chen R, Sun K, Li M, Gu J, Zhuang G, Wei W. Colorectal cancer burden and trends: Comparison between China and major burden countries in the world. Chin J Cancer Res. 2021 Feb 28;33(1):1-10. doi: 10.21147/j.issn.1000-9604.2021.01.01. PMID 33707923
- [Result] Argiles JM. Cancer-associated malnutrition. Eur J Oncol Nurs. 2005;9 Suppl 2:S39-50. doi: 10.1016/j.ejon.2005.09.006. PMID 16437757
- [Result] Hebuterne X, Lemarie E, Michallet M, de Montreuil CB, Schneider SM, Goldwasser F. Prevalence of malnutrition and current use of nutrition support in patients with cancer. JPEN J Parenter Enteral Nutr. 2014 Feb;38(2):196-204. doi: 10.1177/0148607113502674. PMID 24748626
- [Result] Aaldriks AA, van der Geest LG, Giltay EJ, le Cessie S, Portielje JE, Tanis BC, Nortier JW, Maartense E. Frailty and malnutrition predictive of mortality risk in older patients with advanced colorectal cancer receiving chemotherapy. J Geriatr Oncol. 2013 Jul;4(3):218-26. doi: 10.1016/j.jgo.2013.04.001. Epub 2013 Apr 30. PMID 24070460
- [Result] Seo SH, Kim SE, Kang YK, Ryoo BY, Ryu MH, Jeong JH, Kang SS, Yang M, Lee JE, Sung MK. Association of nutritional status-related indices and chemotherapy-induced adverse events in gastric cancer patients. BMC Cancer. 2016 Nov 18;16(1):900. doi: 10.1186/s12885-016-2934-5. PMID 27863481
- [Result] Gellrich NC, Handschel J, Holtmann H, Kruskemper G. Oral cancer malnutrition impacts weight and quality of life. Nutrients. 2015 Mar 27;7(4):2145-60. doi: 10.3390/nu7042145. PMID 25825828
- [Result] Planas M, Alvarez-Hernandez J, Leon-Sanz M, Celaya-Perez S, Araujo K, Garcia de Lorenzo A; PREDyCES(R) researchers. Prevalence of hospital malnutrition in cancer patients: a sub-analysis of the PREDyCES(R) study. Support Care Cancer. 2016 Jan;24(1):429-435. doi: 10.1007/s00520-015-2813-7. Epub 2015 Jun 23. PMID 26099900
- [Result] Cong MH, Li SL, Cheng GW, Liu JY, Song CX, Deng YB, Shang WH, Yang D, Liu XH, Liu WW, Lu SY, Yu L. An Interdisciplinary Nutrition Support Team Improves Clinical and Hospitalized Outcomes of Esophageal Cancer Patients with Concurrent Chemoradiotherapy. Chin Med J (Engl). 2015 Nov 20;128(22):3003-7. doi: 10.4103/0366-6999.168963. PMID 26608978
- [Result] Muscaritoli M, Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Oldervoll L, Ravasco P, Solheim TS, Strasser F, de van der Schueren M, Preiser JC, Bischoff SC. ESPEN practical guideline: Clinical Nutrition in cancer. Clin Nutr. 2021 May;40(5):2898-2913. doi: 10.1016/j.clnu.2021.02.005. Epub 2021 Mar 15. PMID 33946039
- [Result] Tan S, Meng Q, Jiang Y, Zhuang Q, Xi Q, Xu J, Zhao J, Sui X, Wu G. Impact of oral nutritional supplements in post-discharge patients at nutritional risk following colorectal cancer surgery: A randomised clinical trial. Clin Nutr. 2021 Jan;40(1):47-53. doi: 10.1016/j.clnu.2020.05.038. Epub 2020 Jun 2. PMID 32563599
- [Result] Zietarska M, Krawczyk-Lipiec J, Kraj L, Zaucha R, Malgorzewicz S. Chemotherapy-Related Toxicity, Nutritional Status and Quality of Life in Precachectic Oncologic Patients with, or without, High Protein Nutritional Support. A Prospective, Randomized Study. Nutrients. 2017 Oct 11;9(10):1108. doi: 10.3390/nu9101108. PMID 29019951
- [Result] Matthews CE, Moore SC, Arem H, Cook MB, Trabert B, Hakansson N, Larsson SC, Wolk A, Gapstur SM, Lynch BM, Milne RL, Freedman ND, Huang WY, Berrington de Gonzalez A, Kitahara CM, Linet MS, Shiroma EJ, Sandin S, Patel AV, Lee IM. Amount and Intensity of Leisure-Time Physical Activity and Lower Cancer Risk. J Clin Oncol. 2020 Mar 1;38(7):686-697. doi: 10.1200/JCO.19.02407. Epub 2019 Dec 26. PMID 31877085
- [Result] Prabhu Das I, Baker M, Altice C, Castro KM, Brandys B, Mitchell SA. Outcomes of multidisciplinary treatment planning in US cancer care settings. Cancer. 2018 Sep 15;124(18):3656-3667. doi: 10.1002/cncr.31394. Epub 2018 Sep 14. PMID 30216477
- [Result] Ruff SM, Diaz DA, Pitter KL, Hartwell BC, Pawlik TM. Multidisciplinary management in the treatment of intrahepatic cholangiocarcinoma. CA Cancer J Clin. 2023 Jul-Aug;73(4):346-352. doi: 10.3322/caac.21779. Epub 2023 Apr 12. No abstract available. PMID 37046405
- [Result] Lu Z, Fang Y, Liu C, Zhang X, Xin X, He Y, Cao Y, Jiao X, Sun T, Pang Y, Wang Y, Zhou J, Qi C, Gong J, Wang X, Li J, Tang L, Shen L. Early Interdisciplinary Supportive Care in Patients With Previously Untreated Metastatic Esophagogastric Cancer: A Phase III Randomized Controlled Trial. J Clin Oncol. 2021 Mar 1;39(7):748-756. doi: 10.1200/JCO.20.01254. Epub 2021 Jan 8. PMID 33417481
- [Result] Murphy JL, Munir F, Davey F, Miller L, Cutress R, White R, Lloyd M, Roe J, Granger C, Burden S, Turner L. The provision of nutritional advice and care for cancer patients: a UK national survey of healthcare professionals. Support Care Cancer. 2021 May;29(5):2435-2442. doi: 10.1007/s00520-020-05736-y. Epub 2020 Sep 12. PMID 32918612
- [Result] Brown TE, Banks MD, Hughes BGM, Lin CY, Kenny LM, Bauer JD. Randomised controlled trial of early prophylactic feeding vs standard care in patients with head and neck cancer. Br J Cancer. 2017 Jun 27;117(1):15-24. doi: 10.1038/bjc.2017.138. Epub 2017 May 23. PMID 28535154
- [Result] Ratri DMN, Hamidah KF, Puspitasari AD, Farid M. Video-based health education to support insulin therapy in diabetes mellitus patients. J Public Health Res. 2020 Jul 3;9(2):1849. doi: 10.4081/jphr.2020.1849. eCollection 2020 Jul 3. PMID 32728588
- [Result] Bennell KL, Lawford BJ, Keating C, Brown C, Kasza J, Mackenzie D, Metcalf B, Kimp AJ, Egerton T, Spiers L, Proietto J, Sumithran P, Harris A, Quicke JG, Hinman RS. Comparing Video-Based, Telehealth-Delivered Exercise and Weight Loss Programs With Online Education on Outcomes of Knee Osteoarthritis : A Randomized Trial. Ann Intern Med. 2022 Feb;175(2):198-209. doi: 10.7326/M21-2388. Epub 2021 Nov 30. PMID 34843383
- [Result] Cederholm T, Barazzoni R, Austin P, Ballmer P, Biolo G, Bischoff SC, Compher C, Correia I, Higashiguchi T, Holst M, Jensen GL, Malone A, Muscaritoli M, Nyulasi I, Pirlich M, Rothenberg E, Schindler K, Schneider SM, de van der Schueren MA, Sieber C, Valentini L, Yu JC, Van Gossum A, Singer P. ESPEN guidelines on definitions and terminology of clinical nutrition. Clin Nutr. 2017 Feb;36(1):49-64. doi: 10.1016/j.clnu.2016.09.004. Epub 2016 Sep 14. PMID 27642056
- [Result] Loman BR, Luo M, Baggs GE, Mitchell DC, Nelson JL, Ziegler TR, Deutz NE, Matarese LE; NOURISH Study Group. Specialized High-Protein Oral Nutrition Supplement Improves Home Nutrient Intake of Malnourished Older Adults Without Decreasing Usual Food Intake. JPEN J Parenter Enteral Nutr. 2019 Aug;43(6):794-802. doi: 10.1002/jpen.1467. Epub 2018 Nov 22. PMID 30565718
- [Result] Elia M, Normand C, Laviano A, Norman K. A systematic review of the cost and cost effectiveness of using standard oral nutritional supplements in community and care home settings. Clin Nutr. 2016 Feb;35(1):125-137. doi: 10.1016/j.clnu.2015.07.012. Epub 2015 Jul 30. PMID 26309240
- [Result] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- See also: World Health Organization. Cancer. (accessed May 12, 2023) — https://www.who.int/news-room/fact-sheets/detail/cancer
- See also: World Health Organization. Colorectal Cancer Awareness Month 2022 - IARC n.d (accessed May 13, 2023). — https://www.iarc.who.int/featured-news/colorectal-cancer-awareness-month-2022/

DOCUMENTS (2):
  • Study Protocol (2025-03-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT06219083/Prot_002.pdf
  • Informed Consent Form (2025-03-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT06219083/ICF_003.pdf